CLINICAL TRIAL: NCT03627988
Title: Prospective, Multicentric Study Evaluating the Surgical Treatment by Mastectomy With Immediate Prosthetic Breast Reconstruction in Patients With Breast Cancer and Receiving Adjuvant Therapy by TomoTherapy +/-Chemotherapy.
Acronym: MARTA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18 SEIN 11
Record Dates: First submitted 2018-08-02; First posted 2018-08-14 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Invasive
Keywords: Breast Cancer Invasive; TomoTherapy; Immediate prosthetic breast reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with breast cancer (Experimental)
  Interventions: Other: Patients with invasive breast cancer will receive:

INTERVENTIONS:
Other: Patients with invasive breast cancer will receive: — * Mastectomy with Immediate prosthetic breast reconstruction
  * Adjuvant therapy by TomoTherapy (radiation therapy alone or preceded by chemotherapy).

SUMMARY:
Prospective, multicentric, non-randomized phase II study evaluating the surgical treatment by mastectomy with immediate prosthetic breast reconstruction in patients with breast cancer and receiving adjuvant therapy by TomoTherapy +/-Chemotherapy.

Patients with non-inflammatory and non-metastatic invasive mammary carcinoma will be included in this study.

The study procedure will be a surgical treatment by mastectomy with immediate prosthetic breast reconstruction followed by an adjuvant therapy: TomoTherapy +/-Chemotherapy (radiation therapy alone or preceded by chemotherapy).

The nature of the chemotherapy treatment will be decided according to the standards of each center.

The patients will be followed for the study up to 36 months after the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patient with a non-inflammatory and non-metastatic invasive mammary carcinoma.
3. Indication of mastectomy and immediate prosthetic breast reconstruction.
4. Patient wishing to have an immediate mammary reconstruction with prosthesis.
5. Formal or presumptive pre-operative indication for adjuvant radiotherapy (+/- chemotherapy).
6. OMS ≤ 2.
7. Patient affiliated to a Social Health Insurance in France.
8. Patient must provide written informed consent prior to any study specific procedures.

Exclusion Criteria:

1. Metastatic breast cancer.
2. Bilateral breast cancer.
3. Inflammatory breast cancer (T4d).
4. History of breast cancer within 5 years.
5. Not applicable according to the protocol version N°6 : Previous neoadjuvant treatment for the ongoing disease.
6. Pregnant or breastfeeding women.
7. Any psychological, familial, geographical or sociological condition which does not allow to respect the medical follow-up and/or compliance to study procedure.
8. Patient protected by law.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with successful mastectomy strategy by immediate reconstruction. | 12 months for each patient

SECONDARY OUTCOMES:
Quality of the radiotherapy treatment plan (dosimetry). | 78 months for all patients
Progression-free survival. | 36 months for each patient
Early complications assessed using the National Cancer Institute Common Toxicity Criteria for Adverse Effects (NCI-CTCAE) version 4.03. | 36 months for each patient
Late complications assessed using the National Cancer Institute Common Toxicity Criteria for Adverse Effects (NCI-CTCAE) version 4.03. | 36 months for each patient
Quality of Life assessed using the questionnaire called "Breast-Q". | 36 months for each patient
Cosmetic outcome of treated breast assessed using a questionnaire with a Likert scale. | 36 months for each patient

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Bergonie, Bordeaux
  - Institut Universitaire Du Cancer de Toulouse - Oncopole, Toulouse